CLINICAL TRIAL: NCT04096924
Title: A Randomized Multicenter Comparison Trial to Evaluate the Effectiveness and Safety of the Guidewire for Echo-guided Interventions in Treating ASD
Brief Title: A Prospective Randomized Multicenter Trial of the Guidewire for Echo-guided Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Chief, Department of Structural Heart Disease, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYQ001
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Atrial Septal Defect
Keywords: ASD; Atrial septal defects; amplatzer
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Experimental group is allocated to use novel interventional guidewire for the echocardiography guided percutaneous interventions for ASD.
  Interventions: Device: Guidewire for echo-guided interventions
- Control Group (Active Comparator): Control Group is allocated to use Cook lunderquist guidewire for the echocardiography guided percutaneous interventions for ASD.
  Interventions: Device: Cook lunderquist guidewire

INTERVENTIONS:
Device: Guidewire for echo-guided interventions — Under echocardiography guided treatment of ASD with a novel interventional guidewire
  Arms: Treatment Group
Device: Cook lunderquist guidewire — Subjects with ASD treated with amplatzer using the Cook lunderquist guidewire.
  Arms: Control Group

SUMMARY:
Prospective randomized multicenter trial of about 100 subjects enrolled in 3-5 centers. Patients will be randomized to two groups in equal proportion (50 in each). To precise the function of this device on reducing technical difficulties and conquering learning curves, it is required that the doctor should be able to independently do echo-guided percutaneous interventions and his cases should be more than 20 but less than 100. Experimental group is allocated to use novel interventional guidewire for echocardiography guided percutaneous interventions for ASD, control group will be treated by cook lunderquist guidewire. If echo-guided procedure does not work well, the procedure will be immediately replaced by conventional procedure guided by radiology. To evaluate the effectiveness and safety comprehensively, variables are defined as success rate, duration of procedure, times of arrhythmia, times of misguided to tricuspid valve, cardiac perforation, cardiac tamponed, complications in peripheral vessels etc.

DETAILED DESCRIPTION:
1. This is a prospective blinded randomized multicenter comparison clinical trial followed the design of superiority trial to compare the effectiveness and safety of the guidewire for echo-guided interventions designed by Hangzhou Dexin Medical Technological Company with other similar products.
2. This trial will enroll about 100 subjects from 3-5 centers. Patients will be randomized to two groups in equal proportion (50 in each). Proposal recruiting period is 18 months and follow-up will be performed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. age≥2yrs, diameter of defect≥5 mm, central ASD with increased volume load of right heart.
2. edge of defect is ≥5 mm from coronary sinus, superior and inferior vena cava, and pulmonary vein, and≥7 mm from atrioventricular valve.
3. diameter of atrial septal > left-atrium-side diameter of occlude.
4. participants or guardians who can understand the purpose of this trial and voluntarily participate in and sign the informed consent form.

Exclusion Criteria:

1. Primary atrial septal defect.
2. Sinus venosus atrial septal defects.
3. Accompany with endocarditis or hemorrhagic risks.
4. thrombosis in targeting area or venous thrombosis in inserting site.
5. severe pulmonary artery hypertension generated right-to-left shunt.
6. severe myocardial or valve disease unrelated with ASD.
7. suffered infection diseases or developing infection diseases within 1 month, thrombosis in left atrium or left appendage, part or total anomalous pulmonary venous drainage.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-07 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
success rate | Immediately after treatment
  The primary outcome will be the success rate, which is defined by the principles below:
  1. guidewire can successfully access to left atrium through ASD.
  2. sheath can successfully access to left atrium guided by guidewire and not fall into right atrium after guidewire pullout.
  3. guidewire can be successfully pulled out. The secondary outcome will be duration of procedure, times of arrhythmia, times of misguided to tricuspid valve, cardiac perforation, cardiac tamponed, complications in peripheral vessels.

SECONDARY OUTCOMES:
Incidence of major adverse events(MAE) | 1 month
  MAE definition: Any complications related to devices or surgeries, including but not limited to: death, emergency surgery, severe cardiac tamponade requiring pericardiocentesis or operation, hemorrhage, stroke related to operation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD,Ph.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (3):
- China (3):
  - Structural Heart Disease Center, Fuwai Hospital, Beijing, Beijing Municipality
  - Fuwai Huazhong Cardiovascular Hospital, Zhengzhou, Henan
  - Xinjiang People's Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong P, Zhao G, Zhang Z, Zhang W, Fan T, Han Y, Pang K, Wang S, Zhang F, Wang W, Hu S, Pan X. Novel Panna Guide Wire Facilitates Percutaneous and Nonfluoroscopic Procedure for Atrial Septal Defect Closure: A Randomized Controlled Trial. Circ Cardiovasc Interv. 2020 Sep;13(9):e009281. doi: 10.1161/CIRCINTERVENTIONS.120.009281. Epub 2020 Aug 27. PMID 32847382